CLINICAL TRIAL: NCT07087210
Title: In Vivo Quantitative Mapping of Mitochondrial Cardiac Membrane Potential in Heart Failure
Acronym: MITOMAP-HF
Status: Active, not recruiting | Type: Observational
Sponsor: Matthieu Pelletier-Galarneau, MD MSc (Other)
Responsible Party: Sponsor-Investigator, Matthieu Pelletier-Galarneau, MD MSc, MD MSc, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Other Study IDs: ICM 2022-3009
Record Dates: First submitted 2025-03-28; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Mitochondrial Function
Keywords: mitochondrial function; positron emission tomography; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Active: engaged in aerobic exercise (running, cycling, or swimming) for at least 3 days per week or 5 hours per week without extensive layoff over the previous 6 months
  Interventions: Other: Positron Emission Tomography (PET)
- Sedentary: ≤1 structured physical activity per week
  Interventions: Other: Positron Emission Tomography (PET)
- HFpEF: Chronic symptomatic HF and LVEF >40% within 12 months before the screening visit (regardless of the imaging modality)
  Interventions: Other: Positron Emission Tomography (PET)

INTERVENTIONS:
Other: Positron Emission Tomography (PET) — 18F-TPP+ PET/CT imaging

SUMMARY:
This research aims to develop a new method to measure how well mitochondria are working using a special imaging technique called PET (positron emission tomography) with a tracer called 18F-TPP+. This tracer helps us visualize and measure mitochondrial function in a non-invasive way.

DETAILED DESCRIPTION:
Our study has three main goals:

1. Measure Mitochondrial Function in Different Groups: The investigators will compare mitochondrial function in three groups: healthy active individuals, sedentary individuals, and heart failure patients. The investigators expect to see higher mitochondrial function in active individuals and lower function in heart failure patients. The investigators will also test the consistency of our measurements.
2. Correlate Mitochondrial Function with Health Indicators: The investigators will see if our mitochondrial function measurements relate to other health markers, such as exercise capacity, heart health, muscle strength, and cognitive function.
3. Improve the Production of the Tracer: The investigators will refine how they make the 18F-TPP+ tracer to make it more efficient and cost-effective for widespread use in research and clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Active participants:

  1. ≥40 years old
  2. LVEF ≥50%
  3. Body Mass Index <35kg/m2
  4. NYHA fuctional class I
  5. Engaged in aerobic exercise (running cycling or swimming) for ≥3 days per week or 5 hours per week without extensive layoff over the previous 6 months
  6. Non-smoker ≥1 year
  7. Fasting glycemia <6.0 mmol/L
  8. HbA1c <5.7%
* Sedentary participants:

  1. ≥40 years old
  2. LVEF ≥50%
  3. Body Mass Index <35kg/m2
  4. NYHA fuctional class
  5. ≤1 structured physical activity per week
  6. Non-smoker ≥1 year
  7. Fasting glycemia <6.0 mmol/L
  8. HbA1c <5.7%
* HFpEF participants:

  1. Chronic symptomatic HF and LVEF >40% within 12 months before the screening visit (regardless of the imaging modality)
  2. One of the following abnormalities:

     1. HF requiring hospitallization and IV diuretics within 12 months of study entry
     2. NTproBNP >150 pg/ml in sinus rhythm
     3. NTproBNP >450 pg/ml in chronic atrial fibrillation

Exclusion Criteria:

* for all participants :

  1. Infiltrative CMP (e.g., cardiac amyloidosis)
  2. Hypertrophic CMP
  3. Dilated CMP
  4. Ischemic CMP with myocardial infarction
  5. Other chronic diseases or medications that may interfere with mitochondrial function
  6. Primary severe valvular disease
  7. Pericardial disease
  8. Pacemaker
  9. Defibrillator
  10. Congenital heart disease
  11. History of cardiac transplant
  12. BMI >45 kg/m2
  13. High resting blood pressure ≥150/90 mmHg
  14. Estimated glomerular filtration rate (eGFR) <50 mL/min/1.73m2
  15. Iodinated contrast allergy
  16. Women of child bearing potential
  17. Pregnancy
  18. Breastfeeding
  19. Inability to undergo the imaging logistics
  20. Any condition that, in the opinion of the investigator, could compromise the participation in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 Active participants
  10 Sedentary participants
  10 HFpEF participants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Average difference of membrane potential (ΔΨT) in sedentary adults vs subjects with Heart Failure with Preserved Ejection Fraction (HFpEF) | Up to 3 months
  Compare membrane potential (ΔΨT) of patients suffering from Heart Failure with Preserved Ejection Fraction (HFpEF) to healthy sedentary adults matched for age and sex.

SECONDARY OUTCOMES:
Average difference of membrane potential (ΔΨT) in active adults vs healthy sedentary adults | Up to 3 months
  Compare membrane potential (ΔΨT) of healthy active adults to healthy sedentary adult matched for age and sex.
Correlation coefficients between membrane potential (ΔΨT) and ECV vs VO2max, grip strength, left ventricular mass, NT-pro-BNP, neurocognitive function, and NYHA functional class. | Up to 5 months
  Evaluate the correlation between membrane potential (ΔΨT) and ECV with clinical biomarkers of HF including VO2max, grip strength, left ventricular mass, NT-pro-BNP, neurocognitive function, and NYHA functional class.
Coefficient of repeatability between membrane potential (ΔΨT) and ECV repeated measurements. | Up to 3 months
  Evaluate the repeatability of in vivo measurements of membrane potential (ΔΨT) and ECV.

OTHER OUTCOMES:
Correlation between in vivo measurements of membrane potential (ΔΨT) and ECV with metabolites reflecting mitochondrial function. | Up to 3 months
  Explore the association between in vivo measurements of membrane potential (ΔΨT) and ECV with metabolites reflecting mitochondrial function.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided